CLINICAL TRIAL: NCT05817331
Title: Qualitative Interviews to Refine and Assess the Importance of Constructs, and Ensure the Readability of Patient, Carer, and Clinician Versions of the Treatment Preference in Myelodysplasia Questionnaire (TPMQ): pTPMQ, cTPMQ, and mTPMQ, Respectively
Brief Title: Refine and Assess the Readability of Patient, Carer, and Clinician Treatment Preference in Myelodysplasia Questionnaire
Acronym: TPMQ
Status: Completed | Type: Observational
Sponsor: Otsuka Australia Pharmaceutical Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 393-419-00045; 2021_PID02858 (Other: Otsuka Australia Pharmaceutical Pty Ltd)
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Myelodysplastic Syndrome (MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient: Patients with MDS
  Interventions: Other: Patient Treatment Preference Myelodysplasia Questionnaire
- Carer: Carers of patients with MDS
  Interventions: Other: Carer Treatment Preference Myelodysplasia Questionnaire
- Clinician: Clinicians who treat MDS
  Interventions: Other: Clinician Treatment Preference Myelodysplasia Questionnaire

INTERVENTIONS:
Other: Carer Treatment Preference Myelodysplasia Questionnaire — Caregiver-reported outcome measure in MDS
  Groups: Carer
Other: Clinician Treatment Preference Myelodysplasia Questionnaire — Clinician-reported outcome measure in MDS
  Groups: Clinician
Other: Patient Treatment Preference Myelodysplasia Questionnaire — Patient-reported outcome measure (PROM) in MDS
  Groups: Patient

SUMMARY:
The primary goal of this study is to use qualitative interviews to elicit and confirm concepts related to treatment preferences and understandability of the pTPMQ, cTPMQ, and mTPMQ. The information gathered will be used to support the appropriateness of the questionnaires as a patient-reported, caregiver-reported and clinician-reported outcome measure (PROM) in the population of interest.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

A. Adult patients with myelodysplastic syndrome meeting any one of the following criteria:

1. They are currently being treated with azacitidine or
2. They have recently been treated with azacitidine or
3. They have been deemed eligible for treatment with azacitidine, but have not yet commenced treatment

B: Primary caregiver of a patient meeting all of the inclusion criteria (i.e. a patient who meets criteria defined above in A).

C. Clinician treating patients meeting all of the inclusion criteria (i.e. treats patients who meet criteria defined above in A).

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

Exclusion Criteria

A. Patients meeting any of the following criteria are excluded:

1. They have lower risk disease (international prognostic scoring system low or intermediate-1 risk)
2. Cognitive or physical impairment of a nature that makes it infeasible for them to effectively participate in a structured interview.
3. Deemed appropriate for stem cell transplantation and are being pre-treated or will be treated with azacitidine
4. They were treated, are being treated, or will be treated with azacitdine as part of a clinical trial
5. They are a relative of an employee of the investigational clinic, sponsor or research organization (e.g., Investigator, Coordinator, Technician, Interviewer).

B. Carers meeting any of the following criteria are excluded:

1. They are a caregiver of a patient who meets any of the exclusion criteria listed above in A
2. They are a relative of an employee of the investigational clinic, sponsor or research organization (e.g., Investigator, Coordinator, Technician, Interviewer).

C. Clinician will be excluded from participating in the study if a relative of an employee of the sponsor or research organization (e.g., Investigator, Coordinator, Technician, Interviewer).

D. Participants who are not fluent in English, or who cannot read or write in English will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with myelodysplasia who are eligible for treatment with azacitidine or are being treated with azacitidine or have been treated with azacitidine, and Primary carers of the patients such as those mentioned above, and Clinicians who treat patients such as those mentioned above
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Validation of the pTPMQ, cTPMQ and mTPMQ | Each participant is interviewed once for approximately 45 - 60 minutes
  Observational qualitative study consisting of interviews with MDS participants. The study endpoints are an assessment of understanding of the questions, response options and directions, as described in the ISPOR patient-reported outcome measure (PROM) guidance.

CONTACTS AND LOCATIONS:
Overall Officials: Anoop K Enjeti, MBBS FRCP FRCPA PhD, Principal Investigator — Calvary Mater Newcastle, Edith Street, Waratah, NSW 2298 Australia
Locations (1):
- Calvary Mater Newcastle, Newcastle, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No